CLINICAL TRIAL: NCT03501914
Title: Mindfulness Based Intervention for Individuals With Intellectual Disabilities and Their Care Givers: A Pilot Trial
Brief Title: A Pilot Trial of Mindfulness Based Intervention Program for People With Intellectual Disabilities in a Low Income Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILLMINDFULNESS001
Record Dates: First submitted 2018-04-05; First posted 2018-04-18 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Intellectual Disability
Keywords: Care givers; Adults; Intellectual Disability; Mindfulness
MeSH Terms: conditions — Intellectual Disability | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Mindfulness based intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Based Intervention (Experimental): Mindfulness principles based manualized intervention will be provided to the participants which is developed by colleagues in Manchester. This intervention will be adapted to be accessible for people having intellectual disability (ID) in Pakistan.Sessions will take place once-weekly for 12 weeks including an initial orientation session. It will include breathing, soles of the feet, body scan, guided meditation, mindful stretching and walking
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — A mindfulness program based on mindfulness-based principles developed by colleagues in Manchester will be adapted to be accessible for people with intellectual disabilities (ID) in Pakistan. This intervention will be translated into Urdu afterwards focus group will be conducted to get the views from people with ID, thei care takers and other stake holders to adapt and culturally modify the program. It will include some mindfulness based exercises i.e.welcome & introduction, exploring senses, its all in the mind, Mindful eating, breathing, soles of the feet, body scan, guided meditation, mindful stretching and walking.

SUMMARY:
The proposed study is a pre-post intervention study to investigate the acceptability and feasibility of a mindfulness based program for people with intellectual disabilities and their caregivers in a low income setting in Pakistan.

DETAILED DESCRIPTION:
In Pakistan, prevalence of intellectual disability is 19.1/1000 severe intellectual disability and 65/1000 for mild level of intellectual disability. Disability not only affects the individual but also the family in general and caretaker specifically.

Several researches proved that parents of children with disabilities experience number of problems related to parenting stress. There is a dire need to develop feasible, cost-effective, community level interventions, that would augment existing healthcare systems.

Mindfulness as a relatively new therapeutic strategy, has not been practiced as far as individuals with intellectual disability are concerned. This study aims to explore the feasibility and acceptability of mindfulness-based strategies for individuals with intellectual disability and their care takers in improving their well-being. A sample of 12 participants will be recruited from rehabilitation centers. The study will be conducted in Karachi. The group intervention will consist of twelve sessions; approx. 90-minutes per session weekly. therapy logswill be used to measure feasibility and acceptability of the intervention and the full Psychological Therapies Outcome Scale - intellectual disabilities (PTOS)-ID (psychological distress and positive well-being scales) will be used as secondary outcome measure. In addition, the positive well-being section of the PTOS-ID will also be administered at session 3 and 6 as an interim measure of well-being.

Baseline assessment will be done following the consent. Post assessments will be conducted at the end of intervention (at 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Able to cope with 90 minute session (with 10 minute break)
* Able to be in a group setting
* Able to get to the location of the group
* Able to attend most sessions
* All abilities welcome (including individuals who may struggle with language comprehension/expression)
* Able to attend with a consistent staff member/carer for all sessions.

Exclusion Criteria:

* Unable to cope with 90 minute session (with 10 minute break)
* Person struggles with proximity of others or bring in a group setting
* If physically unwell (new onset of severe illness)
* Inconsistent staff team/carers supporting person to sessions
* Ongoing experience of trauma or symptoms of Post-Traumatic Stress Disorder

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
sessions log | from start of intervention till end i.e., 12 Weeks
  We aim to determine whether the mindfulness intervention would be feasible to deliver and acceptable to the participants measured through sessions log

SECONDARY OUTCOMES:
Psychological Therapies Outcome Scale for Intellectual Disabilities (PTOS-ID) | Change in scores from Baseline to 12 Weeks
  PTOS-D will be used to assess psychological distress and positive well being of the participants and caregivers. it is a 29 item scale with 16 questions (Measuring Psychological Distress: higher score indicates higher psychological distress) and 11 questions measuring positive well-being: higher scores indicates higher positive well-being. The other two questions: Q-12 and Q-13 does not contribute to the indexes.

CONTACTS AND LOCATIONS:
Locations (1):
- Dar Ul Sakoon, Karachi, Pakistan

REFERENCES:
- [Background] Chapman, M.J., Hare, D.J., Caton, S., Donalds, D., McInnis, E., & Mitchell, D. (2013). The use of mindfulness with people with intellectual disability: A systematic review and narrative analysis. Mindfulness, 4. Doi: 10.1007/s12671-013-0197-7.